CLINICAL TRIAL: NCT04192461
Title: Accuracy of Tooth Guided Immediate Implant Placement at Molar Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdelrhman Tarek Sahry Abdelazim (Other)
Responsible Party: Sponsor-Investigator, Abdelrhman Tarek Sahry Abdelazim, Doctor, member of oral and maxillofacial surgery RCSEd, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tooth guided immediate implant
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Immediate Implant Placement Guided by the Roots of Multiradicular Teeth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tooth guided immediate implant placement group (Experimental)
  Interventions: Procedure: Tooth guided immediate implant placement

INTERVENTIONS:
Procedure: Tooth guided immediate implant placement — The technique of implant insertion consisted of a progressive preparation of the implant site using the anatomy of the root of the multi-radicular mandibular molars to be extracted as a reference and as an aid to engage the inter-radicular septum

SUMMARY:
Introduction: The concept of immediate implant placement has become popular due to reduced trauma and reduced overall treatment time. Removal of molar teeth provides a challenging and intriguing dilemma due to multiple root morphology. In cases of extraction and immediate placement of implants in the molar region, removal of the inter-radicular septum should be avoided to attain initial implant stability at the time of placement, and prevent slipping of the implant into the extraction socket. Following this technique prevents the slippage of the implant and allows the implant to be guided into the inter-radicular septum.

Objectives: To assess the accuracy of implant placement using the remaining roots of multi-radicular mandibular molars, evaluate bone density around implants and implant stability in fresh extracted site.

Materials and Methods: A prospective study was done on 10 patients with badly destructed mandibular molars. The technique of implant insertion consisted of a progressive preparation of the implant site using the anatomy of the root of the multi-radicular mandibular molars to be extracted as a reference and as an aid to engage the inter-radicular septum.

ELIGIBILITY:
Inclusion Criteria:

* Badly destructed mandibular molar teeth.
* Integrity of the roots.
* Bone coverage of 2/3 of the root.
* Sufficient bone volume.
* Adequate interocclusal distance >7mm.
* Adequate amount of keratinized mucosa.
* Age ranging from 20-45 years.
* Medically fit patients.

Exclusion Criteria:

* Unfavorable position of the tooth or remaining roots.
* Molars with Fused roots.
* Root ankylosis.
* Patients with systemic conditions known to affect the periodontal status and healing such as uncontrolled diabetes and osteoporosis.
* Patients receiving chemotherapy or radiotherapy.
* Heavy smokers.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
implant stability quotient | 3 months
  implant stability quotient will be assessed using Osstell device.
Implant position accuracy using cone beam computed tomography | immediately
  Immediate postoperative and a preoperative conebeam CT will be done. The preoperative and postoperative scans will then be over¬lapped using a dedicated algorithm, which will allow the comparison of the virtually planned and the actual implant positions. Three deviation parameters between each planned and placed implant will be measured. All measurements will be performed using Mimics Innovation Suite 19 ™ software (Materialise Mimics software 3D Medical Imaging, Belgium).
  For analyzing the accuracy, the planned position of the implant will be compared with the actual position of the implant after insertion. Several measuring points will be measured:
  * Horizontal deviation at coronal side of the implant.
  * Horizontal deviation at apex of the implant.
  * Angular deviation.
Bone density around implant | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samraa Elsheikh, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahesh L, Kurtzman GM, Schwartz D, Shukla S. Residual Roots as an Anatomical Guide for Implant Placement: Case Series With Two-Year Follow-up. J Oral Implantol. 2016 Jun;42(3):285-8. doi: 10.1563/aaid-joi-D-15-00101. Epub 2015 Sep 21. PMID 26389698
- [Background] Rodriguez-Tizcareno MH, Bravo-Flores C. Anatomically guided implant site preparation technique at molar sites. Implant Dent. 2009 Oct;18(5):393-401. doi: 10.1097/ID.0b013e3181b4b205. PMID 22129957